CLINICAL TRIAL: NCT01166776
Title: Decellularization of Umbilical Cord Wharton's Jelly for Tissue Regenerative Applications Including Avascular Necrosis
Brief Title: A Research Study Looking at Specific Tissue of the Umbilical Cord
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 12129
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Varices of Umbilical Cord
Keywords: Wharton's jelly; umbilical cord; decellularization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — umbilical cord tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Umbilical cord: To isolate Umbilical cord Wharton's jelly matrix to be used as a scaffold for tissue regenerative applications, including avascular necrosis.

SUMMARY:
The purpose of this study is to isolate Umbilical cord Wharton's jelly matrix to be used as a scaffold for tissue regenerative applications, including avascular necrosis.

DETAILED DESCRIPTION:
Our working hypothesis is that umbilical cord blood Wharton's Jelly matrix has all the biochemical and biomechanical characteristics needed in an ideal scaffold for tissue engineering. Accordingly, we expect matrix to support the growth and differentiation of transplanted mesenchymal stem cells. The first step in this effort is to isolate Wharton's Jelly matrix by decellularization. The second step will be to test the ability of this matrix to support the growth and differentiation of transplanted mesenchymal stem cells. The third step will be to pursue preliminary animal testing to study the ability of this matrix to support bone tissue regeneration in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women
* 18 years of age or older
* willing to donate umbilical cord units

Exclusion Criteria:

* less than 18 years of age
* Has Hepatitis or HIV
* Considered High Risk
* Scheduled for C-Section due to complications during current pregnancy
* Delivered prior to Full Term

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women at time of delivery
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Isolation and decellularization of umbilical cord Wharton's jelly matrix | Immediately upon delivery
  Use the Wharton's Jelly matrix as a scaffold, we should be able to remove the cellular components of Wharton's Jelly. This decellularization process will help decrease antigenicity and accordingly avoid allosensitization. Additionally, the matrix should be able to provide a 3 dimensional (3D) environment needed for biologic and geometric recellularization.

SECONDARY OUTCOMES:
Study the ability of the isolated and decellularized matrix to support recellularization with mesenchymal stem cells and to support their growth and differentiation | Within 24 hours
  Use the decellularized matrix for tissue regeneration purposes, it should be able to support recellularization with undifferentiated mesenchymal stem cells and help support their differentiation into different tissues, including bone or cartilage.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Aljitawi, MD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Children's Mercy Hospital, Kansas City, Missouri